CLINICAL TRIAL: NCT02448836
Title: Deep Transcranial Magnetic Stimulation (dTMS) for the Treatment of Premenstrual Dysphoric Disorder (PMDD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-15-OT-0034-CTIL
Record Dates: First submitted 2015-05-03; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active dTMS treatment (Experimental): In each menstrual cycle, patients will undergo 8 sessions of dTMS active treatment for two weeks (4 sessions every week) with dTMS H-coil system:magstim stimulator rapid2,BrainswayH1coil. The post ovulation phase is the luteal and symptomatic phase of PMDD patients.
  Interventions: Device: dTMS H-coil system:magstim stimulator rapid2,BrainswayH1coil
- Sham dTMS treatment (Sham Comparator): In each menstrual cycle, patients will undergo 8 sessions of Sham dTMS treatment for two weeks (4 sessions every week) with dTMS H-coil system:magstim stimulator rapid2,BrainswayH1coil. The post ovulation phase is the luteal and symptomatic phase of PMDD patients.
  Interventions: Device: Sham: dTMS H-coil system:magstim stimulator rapid2,BrainswayH1coil

INTERVENTIONS:
Device: dTMS H-coil system:magstim stimulator rapid2,BrainswayH1coil — Patients will undergo 8 sessions of dTMS treatment for two weeks (4 sessions every week).
  Arms: Active dTMS treatment
Device: Sham: dTMS H-coil system:magstim stimulator rapid2,BrainswayH1coil — Patients will undergo 8 sessions of Sham dTMS treatment for two weeks (4 sessions every week).
  Arms: Sham dTMS treatment

SUMMARY:
Premenstrual dysphoric disorder (PMDD) is a hormone-dependent mental condition that causes significant suffering in 5% of women of reproductive age worldwide. The prominent symptoms are depressed mood, irritability, mood lability and anxiety. Treatment options for PMDD are limited, with 40% non-responders.

Deep transcranial magnetic stimulation (dTMS) is a novel therapeutic technique, which is based on modulating neural activity by inducing an electric field in the brain. To date, dTMS was found to be an effective treatment for depression, which is highly comorbid with PMDD.

The investigators propose to study the effect of dTMS on PMDD patients in a prospective treatment study.

DETAILED DESCRIPTION:
Premenstrual dysphoric disorder (PMDD) is a hormone-dependent mental condition that causes significant distress in 5% of reproductive age women worldwide. The disorder was recently added to the diagnostic and statistical manual of mental disorders (DSM-5) as one of the mood disorders. PMDD is characterized by affective, cognitive, behavioral, and somatic symptoms. Treatment possibilities are limited, and 30-40% of patients who do not respond to antidepressants or oral contraceptives, are faced with no alternative effective treatment options. PMDD is highly comorbid with major depressive disorder (MDD) and neuroimaging studies in both disorders demonstrate dysfunction of the dorsolateral prefrontal cortex (DLPFC).

Deep transcranial magnetic stimulation (dTMS) is a technique of neuromodulation based on specific anatomic induction of an electric field in the brain. To date, dTMS was proved as an effective treatment tool in a number of mental conditions including drug-resistant major depression, in which the onset of the salutary effect of dTMS was relatively quick (compared with conventional antidepressants). Most clinical trials studying the effect of dTMS in major depression, focused on stimulating the DLPFC.

The investigators propose to conduct a prospective double blind cross-over study, to study the effect of short-term dTMS treatment on PMDD patients.

The aim of this study is to conduct the first evaluation of deep transcranial magnetic stimulation (dTMS) as a treatment option for premenstrual dysphoric disorder (PMDD). The treatment of this recurrent episodic disorder, that effects young, reproductive-age women, poses a significant clinical challenge, as current treatment options imply reproductive impairment (oral contraceptives or GnRH (gonadotropin-releasing hormone) agonists) or disturbing side effects (e.g. sexual side effects in SSRI's (selective serotonin reuptake inhibitor)).

In addition, as many as 40% of women with PMDD do not respond to conventional antidepressants or oral contraceptives, and remain without an effective and tolerable treatment option.

The symptoms of PMDD are episodic and time-limited, and indeed, some of the pharmacological treatment strategies for PMDD consist of intermittent therapy. Thus, he investigators assume that dTMS administered during the 7-14 symptomatic days (after ovulation), may provide a highly needed, tolerable and efficient treatment option for women suffering from this disorder, and may actually prevent the onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

Women at reproductive age (18-50) with a regular menstrual cycle who:

1. Fulfill screening criteria of the premenstrual screening Tool (PSST) for PMDD (Steiner et al., 2003).
2. Report of at least a one year history of regularly experiencing PMDD symptoms, and meet diagnostic criteria for PMDD according to DSM-5 criteria on a clinical psychiatric interview (American Psychiatric Association, 2013).
3. Fulfill criteria for PMDD prospectively, using the daily record of severity of problems (DRSP) (Endicott et al., 2006) for at least two full menstrual cycles of daily symptom charting, by e-mail via a specific software for Internet questionnaires ("Qaultrics"). A cycle will be considered symptomatic if the luteal phase mean score will be 50% greater than the mean follicular phase score (Endicott et al. 2006).
4. Women receiving oral contraceptives (OC) will be included if usage of OC commenced 3 months prior to their enrollment.

Exclusion Criteria:

1. Current pregnancy or getting pregnant during the study.
2. Moderate-severe polycystic ovary syndrome
3. Usage of hormonal IUD (intrauterine device)
4. Recent initiation (less than 3 months) of antidepressant pharmacological treatment.
5. Meet axis I DSM-5 diagnosis for a current major depressive episode or a psychotic disorder at admission.
6. Substance dependence or abuse other than nicotine in the 30 days prior to screening.
7. A personal history of seizures or epilepsy, a history of seizures or epilepsy in first degree relatives and the presence of any known factor that can lower the seizure threshold.
8. Previous head injury and the presence of metallic implants in the cephalic region treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
PMDD symptoms as measured by the PMTS (Premenstrual Tension Syndrome) scales | Patients will be psychiatrically evaluated to assess their mental state and treatment progress throughout the duration of treatments sessions and up to 2 weeks after, an avarage of 6 weeks

SECONDARY OUTCOMES:
PMDD symptoms as measured by DRSP (Daily Record of Severity of Problems) scale | Patients will be psychiatrically evaluated to assess their mental state and treatment progress throughout the duration of treatments sessions and up to 2 weeks after, an avarage of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oren Tene, M.D, Principal Investigator — TASMC Israel